CLINICAL TRIAL: NCT01939613
Title: Colloid Improves Organ Function by Reducing the Elevation of Intra-abdominal Pressure in Resuscitation of Critical Burn Patients
Brief Title: Colloid Improves Organs Function in Resuscitation of Extensive Burn Patients
Status: Completed | Type: Observational
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Principal Investigator, Honghui Zhang, Mr Honghui Zhang, Tang-Du Hospital
Other Study IDs: TDLL-20100180
Record Dates: First submitted 2013-08-30; First posted 2013-09-11 (Estimated); Last update posted 2013-09-11 (Estimated); Status verified 2013-09

CONDITIONS: Burn
Keywords: fluid resuscitation; burn; colloid,; multiple organ dysfunction; intra-abdominal pressure
MeSH Terms: conditions — Burns | interventions — Colloids

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Parkland group: Extensive burn patients are resuscitated with Parkland formula.In the first 24h of resuscitation,crystalloids were infused as the main fluid.
- TMMU group: Extensive burn patients are resuscitated with Third Military Medical University (TMMU) formula as a modified EVANS formula routinely used in China. In the first 24h of resuscitation, crystalloids and colloids were infused together.
  Interventions: Drug: colloids

INTERVENTIONS:
Drug: colloids — TMMU group allows for administration of colloids early,while Parkland group infuse colloids 24 h after burn injury.
  Other Names: frozen fresh plasma
  Groups: TMMU group

SUMMARY:
The present study was to evaluate the effectiveness of colloid compared with crystalloids for fluid resuscitation in critical burn patients with total burn surface area ≥50%.

DETAILED DESCRIPTION:
Extensive burn patients are some of the most challenging critically ill patients who may have multiple-system organ failure with life-threatening complications.Over time, several resuscitation formulae have been proposed to guide burn resuscitation and the best known ones are Parkland and Evans formulae. The main controversy between the two formulae also focuses on whether to infuse the colloid in the first 24 h.Controversy continues and the conflicting results left many clinicians unsure about the effect of colloids on fluid resuscitation in extensive burn patients who suffer higher risk of hypovolaemia, abdominal compartment syndrome (ACS), multiple organs dysfunction and mortality. To address this uncertainty, we conducted a prospective, randomized, controlled clinical trial to compare fluid resuscitation in extensive burns guided by Parkland formulae with TMMU formulae as a modified Evans formula routinely used in China.

ELIGIBILITY:
Inclusion Criteria:

* burn patients with total burn surface area ≥50% and full thickness burn surface area ≥30%.

Exclusion Criteria:

* age <18 yrs, time between burn injury and fluid infusion > 4 h, time arriving at our burn centre > 6 h, pre-existing medical illnesses compromising the cardiopulmonary reserve or those need for compassionate care only.

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: This study was performed in the Department of Burn Intensive Care of the Tangdu Hospital, an academic hospital of the Fourth Military Medical University of Xi'an. populaitons were extensive burns who admitted to our hospital within 4 h since burn injury.
Sampling Method: Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2010-07; Primary Completion 2013-06 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Multiple organs function score (MODS) of extensive burns | 48 hours during fluid resuscitation

SECONDARY OUTCOMES:
Intra-abdominal pressure (IAP) of extensive burns | 48 hours during fluid resuscitation

CONTACTS AND LOCATIONS:
Overall Officials: Xueyong Li, MD, Study Director — Department of Burn and Plastic Sugery
Locations (1):
- Department of Burn and Plastic Surgery,Tangdu Hospital, Xi'an, Shaanxi, China